CLINICAL TRIAL: NCT02328664
Title: The Sensitivity of Scar-biopsies for Residual Colorectal Adenocarcinoma After Endoscopic Resection With Uncertain Radicality
Brief Title: SCar-biopsies After Malignant Colorectal Polypectomy of Uncertain RAdicality
Acronym: SCAPURA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed no added value of second look endoscopy
Sponsor: Dr. Frank ter Borg MD PhD (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other)
Responsible Party: Sponsor-Investigator, Dr. Frank ter Borg MD PhD, MD PhD, Gastroenterologist, Deventer Ziekenhuis
Organization: Deventer Ziekenhuis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCAPURA-Study
Record Dates: First submitted 2014-12-15; First posted 2014-12-31 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer
Keywords: Endoscopic resection; Pathology; Rescue surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flexible sigmoidoscopy or colonoscopy (Other): Subjects will undergo these investigation to take biopsies from the polypectomy scar.
  Interventions: Procedure: Flexible sigmoidoscopy or colonoscopy

INTERVENTIONS:
Procedure: Flexible sigmoidoscopy or colonoscopy — Depending on the localization of the scar of the malignant polyp, either a flexible sigmoidoscopy or colonoscopy will be done to take biopsies from the polypectomy scar.

SUMMARY:
After endoscopic removal of a colorectal polyp that harbors (unexpected) adenocarcinoma, pathology usually can not guarantee a radical resection from an oncological point of view. In such case, additional surgical resection is advised. However, only in 15% of patients, residual adenocarcinoma is found. This study investigates the sensitivity of biopsies from the polypectomy scar for residual adenocarcinoma.

DETAILED DESCRIPTION:
Rationale: colorectal polyps may harbor adenocarcinoma. Numbers are increasing due to the nationwide colorectal screening program. After endoscopic removal, rescue surgery is often performed because radicality can not be guaranteed by the pathologist. However, in 85% of surgical specimen no residual malignancy is found. Given morbidity and mortality associated with surgery a method to diagnose residual cancer is needed.

Biopsies from the polypectomy site are variably used to reduce the likelihood of residual tumor at the polypectomy site under these circumstances. However, the sensitivity of such biopsies is unknown.

Objective: to evaluate the sensitivity of second-look endoscopic biopsies from the polypectomy site for residual tumor.

Study design: prospective cross-sectional design using a multi-center approach. Study population: patients planned for rescue surgery for the sole reason of (potentially) irradical endoscopic resection of a colorectal adenocarcinoma without poor differentiation, lymphovascular invasion or tumor budding and without other signs of dissemination.

Intervention: endoscopic biopsies from the polypectomy site before operation. Main study parameters/endpoints: sensitivity of second-look biopsies from the polypectomy site for residual tumor in the resected bowel and postoperative mortality. Various other factors will be assessed that might be associated with residual cancer.

Nature and extent of the burden and risks associated with participation and benefit: Depending on the situation: a): In case a tattoo needs to be done of the polypectomy site, a second endoscopy is done anyway and taking biopsies (painless) will be of no extra burden; b): In case no tattoo needs to be done a sigmoidoscopy (lesion distal to the splenic flexure) or colonoscopy (proximal to the splenic flexure) needs to be arranged for the purpose of this study. A sigmoidoscopy takes 10-20 minutes. Preparation consists of two enemas. A colonoscopy takes 20-30 minutes. Preparation consists of drinking 3 litre of MoviPrep®, both usually doe at home. Notice that the patient has recent experience with colonoscopy. If necessary, both investigations can be arranged under conscious sedation (the rule in colonoscopy), which also implies day-care admission. The risk of complications of a second endoscopy is estimated < 1:5000. The benefit of a 2nd colonoscopy is the discovery of new polyps in 10-25% of cases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above.
* Endoscopically removed colorectal lesion with the following pathological characteristics:

  * A moderately-to-well differentiated adenocarcinoma.
  * If possible to judge: distance between adenocarcinoma and vertical or lateral resection margin is less than 1 mm.
  * In case of piecemeal resection: unjudgeable radicality (mostly due to loss of orientation and multiple fragments).
  * Absence of / unjudgeable lymphatic / vascular invasion.
  * No or only grade I tumor budding.
* No suspicion of dissemination on the following investigations: serum carcino-embryonic antigen, a computer tomographic (CT) scan of the abdomen and a chest X-ray; in case of a rectal tumor (less than 15 cm from the anal verge): an additional magnetic resonance imaging of the rectum.
* Operation is advised in agreement with the Dutch Guideline on Colorectal cancer, planned and agreed on by the patient.
* Written informed consent is obtained.

Exclusion Criteria:

* Pathology shows one or more of the following characteristics:

  * A radical en-bloc resection with a free vertical and lateral margin of ≧ 1 mm.
  * A poorly differentiated or signet-cell containing adenocarcinoma.
  * Lymphatic or vascular invasion (if this feature is unjudgeable due to piecemeal resection, no exclusion is done).
  * Tumor budding grade II-III.
* Suspicion of dissemination on investigations as mentioned in the inclusion criteria.
* Patients already receiving anti-tumor treatment for another tumor or a synchronic colorectal cancer.
* Patients in whom a second-look endoscopy would require major and unacceptable effort and / or resources, for instance clinical admission for bowel preparation, long travel, general anesthesia, extremely difficult to reach polypectomy site. Such at the decision of the patient and / or treating physician.
* Patient is planned for trans-anal surgery.
* Patient is not planned for surgery.
* Patient is pregnant.
* Patient does not provide written informed consent or is unable to provide such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of biopsies for residual cancer | up to 1 year
  The number of patients with endoscopic biopsies containing adenocarcinoma divided by the number of patients with adenocarcinoma in the resected specimen.

SECONDARY OUTCOMES:
90-day mortality after rescue surgery | 91 days from surgery
  The number of patients that died within 91 day after the operation for presumed residual adenocarcinoma.
The sensitivity of biopsies for residual cancer in the bowel wall | up to 1 year
  The number of patients with endoscopic biopsies containing adenocarcinoma divided by the number of patients with adenocarcinoma in the resected bowel wall (regardless of regional lymph nodes)
The number of complications (defined according to GCP) after biopsies from the polypectomy scar | up to 30 days
  The number of patients with bleeding or perforation after taking biopsies from the polypectomy scar, requiring at least prolongation of treatment, or admission to hospital, or delay or speeding up of surgery.
The sensitivity of global endoscopic assessment of polypectomy site for residual cancer at initial and follow-up endoscopy (to take scar biopsies) | up to 1 year
  The number of patients in whom the endoscopic resection initially and/or at follow-up endoscopic was assessed as incomplete and who also have residual cancer in the surgically resected specimen divided by the total number of patients in whom the endoscopic resection was judged to be incomplete.
The proportion of patients with residual cancer in the resected specimen if malignancy was unsuspected during the endoscopic polypectomy | up to 1 year
  The number of patients in whom the malignancy was initially unsuspected during endoscopic polypectomy and who also have residual cancer in the surgical specimen divided by the total number of patients in whom the malignancy was initially unsuspected during endoscopic polypectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Frank ter Borg, MD PhD, Study Director — Department of Gastroenterology & Hematology, Deventer Hospital
Locations (36):
- Netherlands (36):
  - Medical Center de Veluwe, Apeldoorn, Gelderland
  - Gelre Hospitals, Apeldoorn, Gelderland
  - Hospital Gelderse Vallei, Ede, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Maasstad Hospital Pantein, Beugen, North Brabant
  - Amphia Hospital, Breda, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Bernhoven, Uden, North Brabant
  - The Netherlands Cancer Institute Antoni van Leeuwenhoekhuis, Amsterdam, North Holland
  - Medical Center Slotervaart, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis (Oost & West), Amsterdam, North Holland
  - Academical Medical Center, Gastroenterology department, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Deventer Hospital, Deventer, Overijssel
  - Ziekenhuis Groep Twente, Hengelo, Overijssel
  - Isala Clinics, Zwolle, Overijssel
  - Nij Smellinghe Hospital, Drachten, Provincie Friesland
  - Antonius Hospital Sneek-Emmeloord, Sneek, Provincie Friesland
  - IJsselland Hospital, Capelle aan den IJssel, South Holland
  - Albert Schweitzer Hospital, Dordrecht, South Holland
  - Rivas Zorggroep, Gorinchem, South Holland
  - Groene Hart Hospital, Gouda, South Holland
  - Alrijne Hospital, Leiden, South Holland
  - Erasmus Medical Center, Gastroenterology department, Rotterdam, South Holland
  - Franciscus Gasthuis, Rotterdam, South Holland
  - Maasstad Hospital, Rotterdam, South Holland
  - Ikazia Hospital, Rotterdam, South Holland
  - Vlietland Hospital, Schiedam, South Holland
  - Haga Hospital, The Hague, South Holland
  - Meander Medical Center, Amersfoort, Utrecht
  - Sint Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Groningen, Groningen
  - Martini Hospital, Groningen
  - University Medical Center Utrecht, Gastroenterology department, Utrecht

IPD SHARING:
Plan to Share IPD: No
Data collection is within current OpenClinica standard and not shared

REFERENCES:
- [Background] Mitchell PJ, Haboubi NY. The malignant adenoma: when to operate and when to watch. Surg Endosc. 2008 Jul;22(7):1563-9. doi: 10.1007/s00464-008-9850-y. Epub 2008 Mar 25. PMID 18363065
- [Background] Seitz U, Bohnacker S, Seewald S, Thonke F, Brand B, Braiutigam T, Soehendra N. Is endoscopic polypectomy an adequate therapy for malignant colorectal adenomas? Presentation of 114 patients and review of the literature. Dis Colon Rectum. 2004 Nov;47(11):1789-96; discussion 1796-7. doi: 10.1007/s10350-004-0680-2. PMID 15622570
- [Background] Butte JM, Tang P, Gonen M, Shia J, Schattner M, Nash GM, Temple LK, Weiser MR. Rate of residual disease after complete endoscopic resection of malignant colonic polyp. Dis Colon Rectum. 2012 Feb;55(2):122-7. doi: 10.1097/DCR.0b013e3182336c38. PMID 22228153
- [Background] Meining A, von Delius S, Eames TM, Popp B, Seib HJ, Schmitt W. Risk factors for unfavorable outcomes after endoscopic removal of submucosal invasive colorectal tumors. Clin Gastroenterol Hepatol. 2011 Jul;9(7):590-4. doi: 10.1016/j.cgh.2011.02.002. Epub 2011 Feb 12. PMID 21320641
- [Background] Benizri EI, Bereder JM, Rahili A, Bernard JL, Vanbiervliet G, Filippi J, Hebuterne X, Benchimol D. Additional colectomy after colonoscopic polypectomy for T1 colon cancer: a fine balance between oncologic benefit and operative risk. Int J Colorectal Dis. 2012 Nov;27(11):1473-8. doi: 10.1007/s00384-012-1464-0. Epub 2012 Mar 29. PMID 22454048
- [Background] Di Gregorio C, Bonetti LR, de Gaetani C, Pedroni M, Kaleci S, Ponz de Leon M. Clinical outcome of low- and high-risk malignant colorectal polyps: results of a population-based study and meta-analysis of the available literature. Intern Emerg Med. 2014 Mar;9(2):151-60. doi: 10.1007/s11739-012-0772-2. Epub 2012 Mar 27. PMID 22451095
- [Background] Kitajima K, Fujimori T, Fujii S, Takeda J, Ohkura Y, Kawamata H, Kumamoto T, Ishiguro S, Kato Y, Shimoda T, Iwashita A, Ajioka Y, Watanabe H, Watanabe T, Muto T, Nagasako K. Correlations between lymph node metastasis and depth of submucosal invasion in submucosal invasive colorectal carcinoma: a Japanese collaborative study. J Gastroenterol. 2004 Jun;39(6):534-43. doi: 10.1007/s00535-004-1339-4. PMID 15235870
- [Background] Ueno H, Mochizuki H, Hashiguchi Y, Shimazaki H, Aida S, Hase K, Matsukuma S, Kanai T, Kurihara H, Ozawa K, Yoshimura K, Bekku S. Risk factors for an adverse outcome in early invasive colorectal carcinoma. Gastroenterology. 2004 Aug;127(2):385-94. doi: 10.1053/j.gastro.2004.04.022. PMID 15300569
- [Background] Netzer P, Forster C, Biral R, Ruchti C, Neuweiler J, Stauffer E, Schonegg R, Maurer C, Husler J, Halter F, Schmassmann A. Risk factor assessment of endoscopically removed malignant colorectal polyps. Gut. 1998 Nov;43(5):669-74. doi: 10.1136/gut.43.5.669. PMID 9824349
- [Background] Cooper GS, Xu F, Barnholtz Sloan JS, Koroukian SM, Schluchter MD. Management of malignant colonic polyps: a population-based analysis of colonoscopic polypectomy versus surgery. Cancer. 2012 Feb 1;118(3):651-9. doi: 10.1002/cncr.26340. Epub 2011 Jul 12. PMID 21751204
- [Background] Ikematsu H, Yoda Y, Matsuda T, Yamaguchi Y, Hotta K, Kobayashi N, Fujii T, Oono Y, Sakamoto T, Nakajima T, Takao M, Shinohara T, Murakami Y, Fujimori T, Kaneko K, Saito Y. Long-term outcomes after resection for submucosal invasive colorectal cancers. Gastroenterology. 2013 Mar;144(3):551-9; quiz e14. doi: 10.1053/j.gastro.2012.12.003. Epub 2012 Dec 8. PMID 23232297
- [Derived] Gijsbers KM, Post Z, Schrauwen RWM, Tang TJ, Bisseling TM, Bac DJ, Veenstra RP, Schreuder RM, Epping Stippel LSM, de Vos Tot Nederveen Cappel WH, Slangen RME, van Lelyveld N, Witteman EM, van Milligen de Wit MAWM, Honkoop P, Alderlieste Y, Ter Borg PJC, van Roermund R, Schmittgens S, Dekker E, Leeuwenburgh I, de Ridder RJJ, Zonneveld AM, Hadithi M, van Leerdam ME, Bruno MJ, Vleggaar FP, Moons LMG, Koch AD, Ter Borg F. Low value of second-look endoscopy for detecting residual colorectal cancer after endoscopic removal. Gastrointest Endosc. 2020 Jul;92(1):166-172. doi: 10.1016/j.gie.2020.01.056. Epub 2020 Feb 25. PMID 32105713